CLINICAL TRIAL: NCT01651962
Title: Intravenous Terbutaline to Facilitate Epidural Catheter Placement for Parturients With Labor Pain
Brief Title: Intravenous Terbutaline to Facilitate Labor Epidural Catheter Placement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai Schoenhage (Other)
Responsible Party: Sponsor-Investigator, Kai Schoenhage, Assistant Professor, Anesthesiology Director of Perioperative Services, Director of Liver Transplant Anesthesia, Department of Anesthesiology, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-0412
Record Dates: First submitted 2012-07-20; First posted 2012-07-27 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Labor Pain
Keywords: Labor Pain; Analgesia, Epidural
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Terbutaline; Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Terbutaline (Experimental): Terbutaline 0.125mg i.v. x 1 dose prior to positioning for epidural placement; may repeat x1 PRN
  Interventions: Drug: Terbutaline
- Fentanyl (Active Comparator): Fentanyl 100mcg i.v. x 1 dose prior to positioning for epidural placement; may repeat x1 PRN
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator): 0.9% NaCl i.v. x 1 dose prior to positioning for epidural placement; may repeat x1 PRN
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: Terbutaline
  Arms: Terbutaline
Drug: Fentanyl
  Arms: Fentanyl
Drug: 0.9% NaCl
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Labor pain is a major factor in making the placement of an epidural catheter difficult. The epidural, once in place and dosed, eventually decreases the parturient's pain. To achieve this goal as fast and safely as possible it would be helpful to have a parturient who can tolerate and co-operate with the placement of the epidural catheter.

Briefly stopping contractions, the cause of labor pain, could be the key to achieve this goal.

This study will evaluate the safety, efficacy and duration of the drug terbutaline for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* in labor
* labor pain >3 on visual analog scale (VAS)

Exclusion Criteria:

* cardiovascular disease
* preeclampsia
* diabetes mel-litus
* thyroid disease
* current (outpatient) opioid medication
* recent and / or current use of cocaine
* seizure disorder
* psychiatric disease
* body mass index >35
* preterm labor (<37 weeks pregnant)
* known allergies to any of the three study substances

Ages: 18 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
reduction of pain score on a visual analog scale (VAS) of 1-10 | 0-30 minutes
  semi-quantitative assessment of decrease in the subject's pain score after administration of the study drug for the placement of an epidural catheter

SECONDARY OUTCOMES:
movement during epidural placement | 0-30 minutes
  semi-quantitative assessment of the subject's movement during placement of the epidural catheter: 0-1-2-3: none - extremities - trunk a bit - trunk a lot
position during epidural placement | 0-30 minutes
  semi-quantitative assessment of the subject's position during the epidural catheter placement: 0-1-2: excellent - moderate - poor

OTHER OUTCOMES:
hemodynamic and oxygenation assessment of parturient and fetus, side effects | 0-30 minutes
  heart rate (HR), non-invasive blood pressure (NIBP), pulse-oximetry (SpO2), fetal heart rate (FHR), uterine contractions (CTG - cardiotocogram); feeling of being jittery, pruritus and nausea

CONTACTS AND LOCATIONS:
Overall Officials: Kai Schoenhage, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Tucson Medical Center, Tucson, Arizona
  - University of Arizona Medical Center, Tucson, Arizona